CLINICAL TRIAL: NCT06258629
Title: Resident of Clinical Pathology in Sohag Oncology Center
Brief Title: Prognostic Value of "CD200" in Hematological Malignancies. Hematological Malignancies Comprise a Group of Malignant Clonal Disorders Arising From the Hematopoietic Tissues , Including Leukemia , Multiple Myeloma , and They Have a High Morbidity and Mortality
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reem Yahia Hashim, resident of clinical pathology in sohag oncology center, Sohag University
Other Study IDs: soh-med-24-01-03MS
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group: Age and sex matched healthy control individuals
  Interventions: Diagnostic Test: Flowcytometry on bone marrow aspiration
- Case group: Available number of patients with newly diagnosed as hematological malignancy
  Interventions: Diagnostic Test: Flowcytometry on bone marrow aspiration
- Case group after 6 months: Available number of patients with newly diagnosed as hematological malignancy after 6 months of starting treatment.
  Interventions: Diagnostic Test: Flowcytometry on bone marrow aspiration

INTERVENTIONS:
Diagnostic Test: Flowcytometry on bone marrow aspiration — Flowcytometry on bone marrow aspiration

SUMMARY:
Prognostic value of 'CD200' in hematological malignancies Hematological malignancies comprise a group of malignant clonal disorders arising from the hematopoietic tissues , including leukemia , multiple myeloma , and lymphoma , and they have a high morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed cases of hematological malignancis.

Exclusion Criteria:

* Known cases of hematological malignancies and on treatment.

Ages: 1 Year to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: * Control group of healthy individuals.
  * Newly diagnosed cases of hematological malignancis.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-02-06 (Estimated); Study Completion 2025-02-06 (Estimated)

PRIMARY OUTCOMES:
Level of CD200 diagnostic marker assessed by flow cytometry | one year
  Prognostic value of CD200 in hematological malignancies

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Biondi A, Cazzaniga G. Novel clinical trials for pediatric leukemias: lessons learned from genomic analyses. Hematology Am Soc Hematol Educ Program. 2013;2013:612-9. doi: 10.1182/asheducation-2013.1.612. PMID 24319240
- [Background] Carvajal LA, Neriah DB, Senecal A, Benard L, Thiruthuvanathan V, Yatsenko T, Narayanagari SR, Wheat JC, Todorova TI, Mitchell K, Kenworthy C, Guerlavais V, Annis DA, Bartholdy B, Will B, Anampa JD, Mantzaris I, Aivado M, Singer RH, Coleman RA, Verma A, Steidl U. Dual inhibition of MDMX and MDM2 as a therapeutic strategy in leukemia. Sci Transl Med. 2018 Apr 11;10(436):eaao3003. doi: 10.1126/scitranslmed.aao3003. PMID 29643228
- [Background] Chiaretti S, Vitale A, Cazzaniga G, Orlando SM, Silvestri D, Fazi P, Valsecchi MG, Elia L, Testi AM, Mancini F, Conter V, te Kronnie G, Ferrara F, Di Raimondo F, Tedeschi A, Fioritoni G, Fabbiano F, Meloni G, Specchia G, Pizzolo G, Mandelli F, Guarini A, Basso G, Biondi A, Foa R. Clinico-biological features of 5202 patients with acute lymphoblastic leukemia enrolled in the Italian AIEOP and GIMEMA protocols and stratified in age cohorts. Haematologica. 2013 Nov;98(11):1702-10. doi: 10.3324/haematol.2012.080432. Epub 2013 May 28. PMID 23716539
- [Background] Coles SJ, Wang EC, Man S, Hills RK, Burnett AK, Tonks A, Darley RL. CD200 expression suppresses natural killer cell function and directly inhibits patient anti-tumor response in acute myeloid leukemia. Leukemia. 2011 May;25(5):792-9. doi: 10.1038/leu.2011.1. Epub 2011 Jan 28. PMID 21274000